CLINICAL TRIAL: NCT05667246
Title: Clinical Effect of Caffeine Consumption in Patients Taking Oral Terbinafine
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-03024634
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Terbinafine Adverse Reaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeinated Group (Active Comparator): Caffeinated coffee, 1 cup, 8 oz water setting, 95 mg caffeine
  Interventions: Other: Caffeinated Coffee
- Decaffeinated Group (Placebo Comparator): Decaffeinated coffee, 1 cup, 8 oz water setting
  Interventions: Other: Decaffeinated Coffee

INTERVENTIONS:
Other: Caffeinated Coffee — Subjects would be randomized to a group "Caffeinated" and subjects will be 95 mg of caffeine in caffeinated coffee.
  Arms: Caffeinated Group
Other: Decaffeinated Coffee — Subjects would be randomized to a group "Decaffeinated" and subjects will be no caffeine in decaffeinated coffee.
  Arms: Decaffeinated Group

SUMMARY:
The investigators hypothesize that there would be significant changes in blood pressure or heart rate in patients consuming caffeine while taking terbinafine.

DETAILED DESCRIPTION:
Terbinafine is a common oral medication used for moderate to severe nail onychomycosis. On the terbinafine package insert, it states that terbinafine can reduce clearance of caffeine by 19%. However, the clinical effects of this finding in patients have yet to really be studied. Decreased clearance of caffeine can physically present with measurable signs such as an increased blood pressure or increased heart rate, as well as less measurable symptoms of GI upset, irritability, headache, insomnia. As a result, dermatologists do not always know how to counsel patients taking terbinafine on their caffeine intake. Hence, recommendations vary as no studies have been done on whether caffeine consumption while taking terbinafine is associated with clinical outcomes, such as measurable changes in blood pressure or heart rate.

This will be a preliminary single-blind randomized control clinical study. Patients being started on oral terbinafine by video visit will be approached for enrollment in the study. Patients will be provided with the baseline survey, to assess demographic information, BMI, and daily caffeine intake. Patients with a history of hypertension and anxiety will not be enrolled per the exclusion criteria. If the patient's blood pressure or heart rate are abnormal, they will be removed from the study

We hypothesize that there would be significant changes in blood pressure or heart rate in patients consuming caffeine while taking terbinafine.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any gender at least 18 years of age
* Diagnosed with onychomycosis
* Planning to start oral terbinafine

Exclusion Criteria:

* Pregnant or breastfeeding
* Any history of anxiety or hypertension
* Any patient with an inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | Baseline, 30 min after consuming caffeine, 60 minutes after consuming caffeine
  An inflatable cuff will be placed around the subject's arm. The cuff has a gauge on it that will measure the blood pressure.
Change in Heart Rate | Baseline, 30 min after consuming caffeine, 60 minutes after consuming caffeine
  A heart rate monitor will be used to measure the pulse of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No